CLINICAL TRIAL: NCT03499041
Title: Pharmacokinetics of LY3314814 in Subjects With Hepatic Impairment
Brief Title: A Study of LY3314814 in Participants With Liver Impairment
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Stopped for futility. Phase 3 studies not likely to meet primary endpoints.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16003; I8D-MC-AZEJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3314814 Control (Experimental): LY3314814 administered orally to participants with normal hepatic function
  Interventions: Drug: LY3314814
- LY3314814 Mild (Experimental): LY3314814 administered orally to participants with mild hepatic impairment
  Interventions: Drug: LY3314814
- LY3314814 Moderate (Experimental): LY3314814 administered orally to participants with moderate hepatic impairment
  Interventions: Drug: LY3314814
- LY3314814 Severe (Experimental): LY3314814 administered orally to participants with severe hepatic impairment
  Interventions: Drug: LY3314814

INTERVENTIONS:
Drug: LY3314814 — Administered orally

SUMMARY:
The purpose of the study is to determine whether LY3314814 can be safely prescribed in participants with liver impairment without a dose adjustment. Participants will be on study for 11 days with follow-up about 7 days afterward.

ELIGIBILITY:
Inclusion Criteria:

- Have a Body Mass Index (BMI) of 18 to 40 kilogram per meter square (kg/m²), inclusive, at the time of screening

Exclusion Criteria:

* Have a history of or current significant ophthalmic disease, particularly any eye problem involving the retina
* Have moderate or severe vitiligo or any other clinically significant disorder of skin or hair pigmentation
* Have acute unstable neuropsychiatric disease
* Have active or uncontrolled neurologic disease, or clinically significant head injury

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under The Drug Concentration-Time Curve From Zero To Infinity (AUC[0-∞]) of LY3314814 | Baseline through 240 hours after the administration of study drug
  PK: AUC(0-∞) of LY3314814
PK: Maximum Observed Drug Concentration (Cmax) of LY3314814 | Baseline through 240 hours after the administration of study drug
  PK: Cmax of LY3314814

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Ctr, Orlando, Florida
  - New Orleans Cntr for Clin Res, Knoxville, Tennessee